CLINICAL TRIAL: NCT01656629
Title: Stem Cell Recruitment in Osteoporosis Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to analyze collected samples due to no funds.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NA_00050448
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Low Bone Density
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Teriparatide; Alendronate; Calcium; Vitamin D

ARMS (3):
- teriparatide (Active Comparator): teriparatide 20 mcg sq for 3 months
  Interventions: Drug: Teriparatide
- Alendronate (Active Comparator): 70 mg po weekly for 3 months
  Interventions: Drug: Alendronate
- calcium and vitamin D (Active Comparator): calcium 630 mg vitamin D 500 units daily for 3 months
  Interventions: Dietary Supplement: calcium and vitamin D

INTERVENTIONS:
Drug: Teriparatide — 20 mcg subq daily for 3 months
  Arms: teriparatide
Drug: Alendronate — 70 mg weekly for 3 months
  Arms: Alendronate
Dietary Supplement: calcium and vitamin D
  Arms: calcium and vitamin D

SUMMARY:
Osteoporosis is an important health problem in the rapidly-aging demographic. Fragility fractures are devastating consequences of osteoporosis. The most common treatment approach in osteoporosis is inhibition of bone resorption with drugs like alendronate (ALN). Parathyroid hormone (PTH) stimulates bone formation and is the only anabolic drug available. Dual therapy with ALN and PTH is not as effective as single-drug therapy in preventing fracture. Bone progenitor cells (MSCs) are recruited to sites of bone remodeling when a growth factor called Transforming Growth Factor Beta (TGF-β1) is released from bone. Different osteoporosis medicines may have differing effects on this process. The effects of ALN versus PTH on bone progenitor recruitment in humans are unknown. This is a randomized, clinical trial of ALN, PTH, and calcium and vitamin D in post-menopausal women with low bone mass. Women will be treated for 3 months with ALN or PTH or calcium and vitamin D. Data collected will include bone biopsies for histomorphometry and micro computed tomography (µCT), bone marrow aspirates for molecular studies, peripheral blood to detect circulating bone progenitor cells and dual X-ray absorptiometry. The investigators hypothesize that in humans, PTH will 1) increase bone progenitor number, 2) enhance recruitment of bone progenitor cells to bone resorption sites, and 3) increase bone progenitor number in peripheral circulation. Furthermore, the investigators hypothesize that ALN treatment will have the opposite effect. Understanding the differences in bone progenitor cell activity and recruitment during osteoporosis therapy will provide a mechanistic rationale for effective use of PTH and anti-resorptive drugs in osteoporosis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women aged 50-80 years
* T score < -2.5 at lumbar spine, total hip or femoral neck on dual x-ray absorptiometry (DXA) OR T score < -1.5 with a personal or family history of fracture

Exclusion Criteria:

* Previous use of bisphosphonates or Teriparatide; current estrogen therapy; any other osteoporosis therapy in the past 6 months
* Metabolic bone disease other than osteoporosis
* Body mass index (BMI) < 18
* Weight > 325 lbs
* Current smoking or current alcohol use that exceeds 3 units of alcohol daily
* Use of medications known to affect bone metabolism
* Renal disease, history of kidney stones or hypercalciuria
* Hypo- or hyperparathyroidism; hypo- or hypercalcemia
* Serum vitamin D level < 20 ng/dL
* Refusal to adjust their dietary calcium to <750mg (i.e. two servings per day of calcium rich food)
* History of bone marrow or organ transplant
* History of malignancy or radiation to the bone
* History of esophageal stricture, dysmotility or severe reflux disease
* Gastrointestinal malabsorption
* Use of digoxin
* Need for chronic anticoagulation therapy such as Coumadin, heparin or low molecular weight heparin or inability to discontinue anti-platelet medication
* Bleeding diathesis; hemoglobin ≤ 12.5 g/dL (American Red Cross cut-off to donate blood)
* International normalized ratio (INR) pro time > 1.1 or activated partial thromboplastin time (APT) T ratio > 1.2
* Platelets < 150K/cu mm
* Cellulitis at site of iliac crest
* History of allergy to medications used in bone biopsy (demeclocycline, lidocaine)
* Inability to understand and provide informed consent.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Jan De Beur, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcium and Vitamin D: calcium 630 mg vitamin D 500 units daily for 3 months
  calcium and vitamin D
Period: Overall Study
Arm/Group | Teriparatide | Alendronate | Calcium and Vitamin D
Started | 21 | 18 | 16
Completed | 16 | 16 | 14
Not Completed | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Alendronate | Calcium and Vitamin D | Total
Number analyzed (Participants) | 21 | 18 | 16 | 55
Age, Customized [Count of Participants; unit: Participants]
  18 - 49 years | 0 | 0 | 0 | 0
  50 - 80 years | 21 | 18 | 16 | 55
  81 - 100 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 16 | 55
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 16 | 55

OUTCOME MEASURES:

1. Primary Outcome: The Percent Change in Circulating Osteoprogenitor Cells as Assessed by Flow Cytometry in the Blood Before and After Treatment With Parathyroid Hormone (PTH) or Alendronate (ALN).
Time Frame: up to 3 months
Measure: Mean (Standard Deviation); unit: percent change in osteoprogenitor cells
Arm/Group | Teriparatide | Alendronate | Calcium and Vitamin D
Number analyzed (Participants) | 16 | 16 | 14
percent change in osteoprogenitor cells | 0.0000242 (0.0000283) | 0.0000104 (0.0000231) | -0.0000068 (0.0000449)

2. Secondary Outcome: Difference in Bone Formation as Assessed by Bone Histomorphometry on Bone Biopsy Between Treatment Groups
Time Frame: 3 months
Population: Collected bone biopsy samples were not analyzed and no data was generated. Therefore data was not collected.
Arm/Group | Teriparatide | Alendronate | Calcium and Vitamin D
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Difference in Osteogenic Potential of Bone Marrow as Measure by Colony Forming Unit Osteoblast (CFU-Ob) Assays Between Treatment Groups
Time Frame: 3 months
Population: Collected osteoblast assay samples were not analyzed and no data was generated. Therefore data was not collected.
Arm/Group | Teriparatide | Alendronate | Calcium and Vitamin D
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Each participant was followed for 14 weeks for adverse events
Arm/Group | Teriparatide | Alendronate | Calcium and Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 2/21 | 0/18 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=21) | Alendronate (N=18) | Calcium and Vitamin D (N=16)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There was a high level of variability and this data has not been validated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes